CLINICAL TRIAL: NCT00600366
Title: Efficacy and Safety of Biphasic Insulin Aspart 30 in Insulin Naive Type 2 Diabetic Patients With Secondary OHA Failure
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 FlexPen® in Insulin Naive Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1566
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
  Other Names: BIASP; NovoMix 30; NovoLog 70/30 Mix

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the efficacy of biphasic insulin aspart 30 on blood glucose control in insulin naive type 2 diabetes failing on secondary oral hypoglycaemic agent (OHA).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin naive diabetes
* Current treatment with OHA, secondary failure
* Body mass index (BMI) below 40 kg/m2
* HbA1c over 8.5%
* Willing and able to start with insulin therapy and to perform self-blood glucose monitoring

Exclusion Criteria:

* History of drug or alcohol abuse
* Receipt of the investigational drug within the last month prior to this trial
* Known or suspected allergy to trial products or related products
* Severe uncontrolled hypertension
* Any disease or condition, which the Investigator feels, would interfere with the trial

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2004-03; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 12 weeks of treatment

SECONDARY OUTCOMES:
Blood glucose profiles
Incidence of hypoglycaemic episodes
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Serbia and Montenegro (4):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Nis
  - Novo Nordisk Investigational Site, Novi Sad

REFERENCES:
- [Result] Lalic NM, Micic D, Antic S, Bajovic L, Pantelinac P, Jotic A, Kendereski A, Dimic D, Djukic A, Mitrovic M, Vujasin M. Effect of biphasic insulin aspart on glucose and lipid control in patients with Type 2 diabetes mellitus. Expert Opin Pharmacother. 2007 Dec;8(17):2895-901. doi: 10.1517/14656566.8.17.2895. PMID 18001251
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com